CLINICAL TRIAL: NCT01096160
Title: A Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK-8266
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK8266 in Hypertensive Men (MK-8266-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 8266-002; 2010-018654-13 (EudraCT Number)
Record Dates: First submitted 2010-03-26; First posted 2010-03-30 (Estimated); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-06

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Panel A: MK-8266 BID, 1 mg/Placebo (Experimental): MK-8266 1 mg (0.7 mg in the morning [AM] + 0.3 mg in the evening [PM]), or as matching placebo BID.
  Interventions: Drug: MK-8226 BID, 1 mg; Drug: Placebo BID (Panel A)
- Panel B: MK-8266 BID, 1.8 mg/Placebo (Experimental): MK-8266 1.8 mg (1 mg in the AM + 0.8 mg in the PM), or as matching placebo BID.
  Interventions: Drug: MK-8266 BID, 1.8 mg; Drug: Placebo BID (Panel B)
- Panel C: MK-8266 TID, 1.8 mg/Placebo (Experimental): MK-8266 TID, 1.8 mg (0.6 mg every 6 hours [q6hr]), or as matching placebo TID.
  Interventions: Drug: MK-8266 TID, 1.8 mg; Drug: Placebo TID (Panel C)
- Panel D: MK-8266 TID, 2.4 mg/Placebo (Experimental): MK-8266 TID (Panel D), 2.4 mg (0.8 mg q6hr), or as matching placebo TID. Panel D was completed prior to initiation of Panel E.
  Interventions: Drug: MK-8266 TID, 2.4 mg; Drug: Placebo TID (Panel D)
- Panel E: MK-8266 TID, 2.4 mg/Placebo (Experimental): MK-8266 TID (Panel E), 2.4 mg (0.8 mg q6hr), or as matching placebo TID. Panel E was initiated after completion of Panel D.
  Interventions: Drug: MK-8266 TID, 2.4 mg; Drug: Placebo TID (Panel E)

INTERVENTIONS:
Drug: MK-8226 BID, 1 mg — MK-8266 1 mg administered as oral capsules (0.7 mg + 0.3 mg), BID for 10 consecutive days. Panel A was completed prior to initiation of Panel B.
  Other Names: MK-8266
  Arms: Panel A: MK-8266 BID, 1 mg/Placebo
Drug: MK-8266 BID, 1.8 mg — MK-8266 1.8 mg administered as oral capsules (1 mg + 0.8 mg), BID for 10 consecutive days. Panel B was completed prior to initiation of Panel C.
  Other Names: MK-8266
  Arms: Panel B: MK-8266 BID, 1.8 mg/Placebo
Drug: MK-8266 TID, 1.8 mg — MK-8266 1.8 mg administered as oral capsules (0.6 mg), TID for 10 consecutive days. Panel C was completed prior to initiation of Panel D.
  Other Names: MK-8266
  Arms: Panel C: MK-8266 TID, 1.8 mg/Placebo
Drug: MK-8266 TID, 2.4 mg — MK-8266 TID (Panel D), 2.4 mg administered as oral capsules (0.8 mg), TID for 10 consecutive days. Panel D was completed prior to initiation of Panel E.
  Other Names: MK-8266
  Arms: Panel D: MK-8266 TID, 2.4 mg/Placebo
Drug: MK-8266 TID, 2.4 mg — MK-8266 TID (Panel E), 2.4 mg administered as oral capsules (0.8 mg), TID for 10 consecutive days. Panel E was initiated after completion of Panel D.
  Other Names: MK-8266
  Arms: Panel E: MK-8266 TID, 2.4 mg/Placebo
Drug: Placebo BID (Panel A) — Placebo administered as oral capsules BID for 10 consecutive days. Panel A was completed prior to initiation of Panel B.
  Arms: Panel A: MK-8266 BID, 1 mg/Placebo
Drug: Placebo BID (Panel B) — Placebo administered as oral capsules BID for 10 consecutive days. Panel B was completed prior to initiation of Panel C.
  Arms: Panel B: MK-8266 BID, 1.8 mg/Placebo
Drug: Placebo TID (Panel C) — Placebo administered as oral capsules TID for 10 consecutive days. Panel C was completed prior to initiation of Panel D.
  Arms: Panel C: MK-8266 TID, 1.8 mg/Placebo
Drug: Placebo TID (Panel D) — Placebo administered as oral capsules TID for 10 consecutive days. Panel D was completed prior to initiation of Panel E.
  Arms: Panel D: MK-8266 TID, 2.4 mg/Placebo
Drug: Placebo TID (Panel E) — Placebo administered as oral capsules TID for 10 consecutive days. Panel E was initiated after completion of Panel D.
  Arms: Panel E: MK-8266 TID, 2.4 mg/Placebo

SUMMARY:
This study evaluated adverse events (AEs), study discontinuation due to AEs, and pharmacodynamics of MK-8266 in male participants with mild to moderate hypertension.

DETAILED DESCRIPTION:
This study evaluated AEs, discontinuation due to AEs, and effects on hemodynamic parameters, including systolic blood pressure (SBP) and aortic augmentation index (AIx), following multiple oral doses of MK-8266. Five serial panels, each consisting of eight participants (40 participants in Panels A, B, C, D, and E), were randomized to receive either MK-8266 or matching placebo twice daily (BID) or three times daily (TID) for 10 consecutive days. Although the original plan was to evaluate MK-8266 treatment in Panels D and E using both BID and TID regimens, the study actually evaluated identical TID regimens in these panels.

ELIGIBILITY:
Inclusion Criteria:

* Participant is male with essential hypertension (high blood pressure)
* Participant is in good general health (with the exception of hypertension)
* Participant has a Body Mass Index (BMI) <= 33 kg/m^2 at the Screening visit
* Participant has a platelet count >= 150,000 cu/mL at the Screening visit
* Participant has a positive AIx at the Screening visit

Exclusion Criteria:

* Participant has a history of stroke, chronic seizure, or major neurological disease
* Participant has a functional disability that can interfere with rising from a seated position to the standing position
* Participant has any history of a bleeding or clotting disorder
* Participant has a history of cancer
* Participant is unable to refrain from or anticipates the use of any prescription or non-prescription medication
* Participant consumes excessive amounts of alcohol or caffeinated beverages daily

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2010-11-01 (Actual); Study Completion 2010-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Panel A: MK-8266 BID (1 mg): MK-8266 BID 1 mg, administered as oral capsules (0.7 mg AM + 0.3 mg PM) for 10 days
- Panel A: Placebo BID: Matching placebo capsules, administered orally for 10 days
- Panel B: MK-8266 BID (1.8 mg): MK-8266 BID 1.8 mg, administered as oral capsules (1 mg AM + 0.8 mg PM) for 10 days
- Panel B: Placebo BID: Matching placebo capsules, administered orally BID for 10 days
- Panel C: MK-8266 TID (1.8 mg): MK-8266 0.6 mg TID, administered as oral capsules (1.8 mg) for 10 days
- Panel C: Placebo TID; Panel D: Placebo TID; Panel E: Placebo TID: Matching placebo capsules, administered orally TID for 10 days
- Panel D: MK-8266 TID (2.4 mg); Panel E: MK-8266 TID (2.4 mg): MK-8266 0.8 mg TID, administered as oral capsules (2.4 mg) for 10 days
Period: Overall Study
Arm/Group | Panel A: MK-8266 BID (1 mg) | Panel A: Placebo BID | Panel B: MK-8266 BID (1.8 mg) | Panel B: Placebo BID | Panel C: MK-8266 TID (1.8 mg) | Panel C: Placebo TID | Panel D: MK-8266 TID (2.4 mg) | Panel D: Placebo TID | Panel E: MK-8266 TID (2.4 mg) | Panel E: Placebo TID
Started | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Completed | 6 | 2 | 5 | 2 | 5 | 2 | 4 | 2 | 4 | 1
Not Completed | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Met stopping criteria per protocol | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Panel A: MK-8266 BID, 1 mg: MK-8266 BID 1 mg, administered as oral capsules (0.7 mg AM + 0.3 mg PM) for 10 days, or as matching placebo
- Panel B: MK-8266 BID, 1.8 mg: MK-8266 BID 1 mg, administered as oral capsules (1 mg AM + 0.8 mg PM) for 10 days
- Panel B: Placebo BID; Panel C: Placebo TID; Panel D: Placebo TID; Panel E: Placebo TID: Matching placebo capsules, administered orally for 10 days
- Panel C: MK-8266 TID, 1.8 mg: MK-8266 TID 1.8 mg, administered as oral capsules (0.6 mg q6hr) for 10 days
- Panel D: MK-8266 TID, 2.4 mg; Panel E: MK-8266 TID, 2.4 mg: MK-8266 TID 2.4 mg, administered as oral capsules (0.8 mg q6hr) for 10 days
- Total: Total of all reporting groups
Arm/Group | Panel A: MK-8266 BID, 1 mg | Panel A: Placebo BID | Panel B: MK-8266 BID, 1.8 mg | Panel B: Placebo BID | Panel C: MK-8266 TID, 1.8 mg | Panel C: Placebo TID | Panel D: MK-8266 TID, 2.4 mg | Panel D: Placebo TID | Panel E: MK-8266 TID, 2.4 mg | Panel E: Placebo TID | Total
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (1.5) | 47.5 (4.9) | 45.5 (7.8) | 52.0 (1.4) | 46.5 (3.4) | 54.0 (1.4) | 46.2 (5.5) | 46.5 (7.8) | 47.2 (5.2) | 48.5 (0.7) | 47.6 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 40
Baseline HR [Median (Full Range); unit: Beats per minute] — Measurements of HR were obtained in triplicate using a validated, semi-automated oscillometric device, and the triplicate measurements were recorded as median values Population: All participants who received at least one dose of the investigational drug
  Beats per minute | 70 [53 to 91] | 90 [71 to 108] | 79 [71 to 92] | 89 [79 to 99] | 74 [43 to 85] | 69 [65 to 72] | 72 [59 to 84] | 88 [79 to 96] | 74 [60 to 127] | 81 [67 to 94] | 73 [43 to 127]

OUTCOME MEASURES:

1. Primary Outcome: Participants Receiving MK-8266 or Placebo Who Experienced At Least One Adverse Event (AE) During Treatment and Postdose Follow-up
Description: Assessment of the number of participants with at least one clinical or laboratory AE in those receiving multiple oral doses of MK-8266. An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the sponsor's product, whether or not considered related to the use of the product.
Time Frame: Up to 24 days
Population: All participants who received at least one dose of the investigational drug
Measure: Number; unit: Count of Participants
Groups:
- Panel A: MK-8266 BID (1 mg): MK-8266 1 mg (0.7 mg AM + 0.3 mg PM), administered orally for 10 days
- Panel A: Placebo; Panel B: Placebo: Matching placebo capsules, administered orally BID for 10 days
- Panel B: MK-8266 BID (1.8 mg): MK-8266 1.8 mg (1 mg AM + 0.8 mg PM), administered orally for 10 days
- Panel C: Placebo; Panel D: Placebo; Panel E: Placebo: Matching placebo capsules, administered orally TID for 10 days
Arm/Group | Panel A: MK-8266 BID (1 mg) | Panel A: Placebo | Panel B: MK-8266 BID (1.8 mg) | Panel B: Placebo | Panel C: MK-8266 TID (1.8 mg) | Panel C: Placebo | Panel D: MK-8266 TID (2.4 mg) | Panel D: Placebo | Panel E: MK-8266 TID (2.4 mg) | Panel E: Placebo
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Count of Participants | 5 | 0 | 5 | 1 | 3 | 1 | 4 | 1 | 5 | 2

2. Primary Outcome: Participants Receiving MK-8266 or Placebo Who Discontinued Treatment Due to an AE
Description: Assessment of the number of participants receiving MK-8266 who discontinued therapy due to an AE over 10 days of treatment. An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product. The number of participants in any treatment group who discontinued therapy due to an AE was primarily assessed for Days 0-10.
Time Frame: Up to 10 days
Population: All participants who received at least one dose of the investigational drug
Measure: Number; unit: Count of Participants
Groups:
- Panel C: MK-8266 TID, 1.8 mg: MK-8266 0.6 mg TID as oral capsules (1.8 mg) for 10 days
- Panel E: MK-8266 2.4 mg TID: MK-8266 0.8 mg TID, administered as oral capsules (2.4 mg) for 10 days
Arm/Group | Panel A: MK-8266 BID (1 mg) | Panel A: Placebo | Panel B: MK-8266 BID (1.8 mg) | Panel B: Placebo | Panel C: MK-8266 TID, 1.8 mg | Panel C: Placebo | Panel D: MK-8266 TID (2.4 mg) | Panel D: Placebo | Panel E: MK-8266 2.4 mg TID | Panel E: Placebo
Number analyzed (Participants) | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 6 | 2
Count of Participants | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

3. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) Following Multiple Oral Doses of MK-8266 or Placebo
Description: Assessment of the change from baseline in SBP, obtained using a validated, semi-automated oscillometric device. Evaluated for MK-8266 relative to placebo in participants, as measured by the time weighted average change over 24 hours postdose (TWA^0-24hrs) on dosing Day 10. Panel D and Panel E had identical treatments (MK-8266 0.8 mg TID), which were combined for this analysis.
Time Frame: Baseline and Day 10
Population: All participants who received at least one dose of the investigational drug and had SBP assessments at Baseline and on Day 10
Measure: Least Squares Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Groups:
- Panel A: MK-8266 BID, 1 mg: MK-8266 1 mg (0.7 mg AM + 0.3 mg PM), administered orally for 10 days
- Panel B: MK-8266 BID, 1.8 mg: MK-8266 1.8 mg (1 mg AM+ 0.8 mg PM), administered orally for 10 days
- Panels D & E Combined: MK-8266 TID, 2.4 mg: MK-8266 0.8 mg TID, administered as oral capsules (2.4 mg) for 10 days. Panel D was completed prior to initiation of Panel E.
- Pooled Placebo: Matching placebo capsules from Panels A, B, C, D & E, administered orally BID or TID for 10 days
Arm/Group | Panel A: MK-8266 BID, 1 mg | Panel B: MK-8266 BID, 1.8 mg | Panel C: MK-8266 TID, 1.8 mg | Panels D & E Combined: MK-8266 TID, 2.4 mg | Pooled Placebo
Number analyzed (Participants) | 6 | 5 | 5 | 8 | 9
Millimeters of mercury (mmHg)
  Baseline value | 141.5 (8.96) | 132.6 (6.66) | 148.6 (23.77) | 134.5 (8.98) | 146.7 (12.07)
  Change from Baseline at Day 10 | -5.09 (7.04) | -2.18 (6.80) | -4.78 (7.64) | 0.77 (6.62) | -3.18 (7.72)
Statistical Analysis 1: Comparison: Panel A: MK-8266 BID, 1 mg vs Pooled Placebo; Test type: Other — Difference in change from baseline in SBP (TWA^0-24hrs); p = 0.1194, Linear mixed effects model; Mean Difference (Final Values) = -7.08, 90% CI 2-sided [-17.1 to 2.92]
Statistical Analysis 2: Comparison: Panel B: MK-8266 BID, 1.8 mg vs Pooled Placebo; Test type: Other — Difference in change from baseline in SBP (TWA^0-24hrs); p = 0.0224, Linear mixed effects model; Mean Difference (Final Values) = -13.1, 90% CI 2-sided [-23.7 to -2.48]
Statistical Analysis 3: Comparison: Panel C: MK-8266 TID, 1.8 mg vs Pooled Placebo; Test type: Other — Difference in change from baseline in SBP (TWA^0-24hrs); p = 0.4791, Linear mixed effects model; Mean Difference (Final Values) = 0.33, 90% CI 2-sided [-10.3 to 10.91]
Statistical Analysis 4: Comparison: Panels D & E Combined: MK-8266 TID, 2.4 mg vs Pooled Placebo; Panel D and Panel E had identical treatments (MK-8266 0.8 mg TID), which were combined for this analysis. Panel D was completed prior to initiation of Panel E; Test type: Other — Difference in change from baseline in SBP (TWA^0-24hrs); p = 0.0705, Linear mixed effcts model; Mean Difference (Final Values) = -8.21, 90% CI 2-sided [-17.4 to 1.01]

4. Primary Outcome: Heart Rate (HR) on Day 10 Following Multiple Oral Doses of MK-8266 or Placebo
Description: Assessment of HR (beats/min) on Day 10 (24-hours postdose) with MK-8266 relative to placebo in participants, as measured by the time weighted average change over 24 hours postdose (TWA^0-24hrs). Panel D and Panel E had identical treatments (MK-8266 0.8 mg TID), which were combined for this analysis. Baseline HR values are shown in the Baseline Characteristics section for Panels A, B, C, D, E.
Time Frame: Day 10 (24 hours postdose)
Population: All participants who received at least one dose of the investigational drug and had HR assessments 24 hours postdose on Day 10.
Measure: Mean (Standard Deviation); unit: Beats per minute
Groups:
- Panels D & E Combined: MK-8266 TID: MK-8266 TID (2.4 mg): MK-8266 0.8 mg TID, administered as oral capsules (2.4 mg) for 10 days. Panel D was completed prior to initiation of Panel E.
- Pooled Placebo: Matching placebo capsules, administered orally TID for 10 days
Arm/Group | Panel A: MK-8266 BID (1 mg) | Panel B: MK-8266 BID (1.8 mg) | Panel C: MK-8266 TID (1.8 mg) | Panels D & E Combined: MK-8266 TID: MK-8266 TID (2.4 mg) | Pooled Placebo
Number analyzed (Participants) | 6 | 5 | 5 | 8 | 9
Beats per minute | 65.89 (5.59) | 69.32 (7.87) | 62.30 (5.28) | 66.10 (5.38) | 62.04 (5.98)
Statistical Analysis 1: Comparison: Panel A: MK-8266 BID (1 mg) vs Pooled Placebo; Test type: Other — Comparison of Day 10 values (TWA^0-24hrs) for MK-8266 vs placebo; p = 0.1161, Linear mixed effects model; Mean Difference (Final Values) = 3.85, 90% CI 2-sided [-1.51 to 9.22]
Statistical Analysis 2: Comparison: Panel B: MK-8266 BID (1.8 mg) vs Pooled Placebo; Test type: Other — Comparison of Day 10 values (TWA^0-24hrs) for MK-8266 vs placebo; p = 0.0189, Linear mixed effects model; Mean Difference (Final Values) = 7.28, 90% CI 2-sided [1.60 to 12.97]
Statistical Analysis 3: Comparison: Panel C: MK-8266 TID (1.8 mg) vs Pooled Placebo; Test type: Other — Comparison of Day 10 values (TWA^0-24hrs) for MK-8266 vs placebo; p = 0.4689, Linear mixed effects model; Mean Difference (Final Values) = 0.26, 90% CI 2-sided [-5.42 to 5.95]
Statistical Analysis 4: Comparison: Panels D & E Combined: MK-8266 TID: MK-8266 TID (2.4 mg) vs Pooled Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Other — Comparison of Day 10 values (TWA^0-24hrs) for MK-8266 vs placebo; p = 0.0869, Linear mixed effects model; Mean Difference (Final Values) = 4.06, 90% CI 2-sided [-0.89 to 9.01]

5. Secondary Outcome: Aortic Augmentation Index (AIx) on Day 10 Following Multiple Oral Doses of MK-8266 or Placebo
Description: Assessment of the central, ascending aortic blood pressure augmentation index (AIx), based on measurement of central pulse pressure at selected time points on Day 10, as measured by applanation tonometry of the radial artery. This outcome measure assessed the time weighted average change over 24 hours postdose (TWA^0-24hrs) on dosing Day 10. Panel D and Panel E had identical treatments (MK-8266 0.8 mg TID), which were combined for this assessment.
Time Frame: Day 10
Population: All participants who received at least one dose of the investigational drug and had AIx assessment on Day 10
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | Panel A: MK-8266 BID, 1 mg | Panel B: MK-8266 BID, 1.8 mg | Panel C: MK-8266 TID, 1.8 mg | Panels D & E Combined: MK-8266 TID, 2.4 mg | Pooled Placebo
Number analyzed (Participants) | 6 | 5 | 5 | 8 | 9
mmHg | 8.81 (4.86) | 7.45 (2.59) | 13.50 (8.95) | 11.89 (7.00) | 18.68 (6.68)
Statistical Analysis 1: Comparison: Panel A: MK-8266 BID, 1 mg vs Pooled Placebo; Test type: Other — Comparison of Day 10 values (TWA^0-24hrs) for MK-8266 vs placebo; p = 0.003, Linear mixed effects model; Mean Difference (Final Values) = -9.87, 90% CI 2-sided [-15.7 to -4.09]
Statistical Analysis 2: Comparison: Panel B: MK-8266 BID, 1.8 mg vs Pooled Placebo; Test type: Other — Comparison of Day 10 values (TWA^0-24hrs) for MK-8266 vs placebo; p = 0.002, Linear mixed effects model; Mean Difference (Final Values) = -11.2, 90% CI 2-sided [-17.3 to -5.10]
Statistical Analysis 3: Comparison: Panel C: MK-8266 TID, 1.8 mg vs Pooled Placebo; Test type: Other — Comparison of Day 10 values (TWA^0-24hrs) for MK-8266 vs placebo; p = 0.080, Linear mixed effcts model; Mean Difference (Final Values) = -5.18, 90% CI 2-sided [-11.3 to 0.95]
Statistical Analysis 4: Comparison: Panels D & E Combined: MK-8266 TID, 2.4 mg vs Pooled Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Other — Difference in change from baseline in AIx (TWA^0-24hrs); p = 0.019, Linear mixed effcts model; Mean Difference (Final Values) = -6.79, 90% CI 2-sided [-12.1 to -1.46]

6. Secondary Outcome: Change From Baseline in Cyclic Guanosine Monophosphate (cGMP) Following Multiple Oral Doses of MK-8266 or Placebo
Description: Assessment of whole blood samples for cGMP analysis, based on samples obtained predose as well as 4 and 24 hours postdose on Day 1 and Day 10, and predose only on Day 4. The change from baseline in cGMP was assessed at 24 hours postdose on Day 10. Panel D and Panel E had identical treatments (MK-8266 0.8 mg TID), which were combined for this assessment.
Time Frame: Baseline and Day 10
Population: All participants who received at least one dose of the investigational drug and had cGMP assessments at Baseline and on Day 10
Measure: Least Squares Mean (Standard Deviation); unit: nanomoles (nM)
Arm/Group | Panel A: MK-8266 BID, 1 mg | Panel B: MK-8266 BID, 1.8 mg | Panel C: MK-8266 TID, 1.8 mg | Panels D & E Combined: MK-8266 TID, 2.4 mg | Pooled Placebo
Number analyzed (Participants) | 6 | 5 | 5 | 8 | 9
nanomoles (nM)
  Baseline value | 1.61 (0.77) | 0.74 (0.50) | 1.69 (1.15) | 2.68 (1.29) | 0.54 (0.21)
  Change from Baseline at Day 10 | 1.34 (2.74) | 1.74 (4.62) | 0.43 (0.66) | 0.81 (2.78) | 1.05 (1.16)
Statistical Analysis 1: Comparison: Panel A: MK-8266 BID, 1 mg vs Pooled Placebo; Test type: Other — Difference in change from baseline in cGMP; p = 0.318, Linear mixed effects model; Geometric Mean Ratio = 1.28, 90% CI 2-sided [0.53 to 3.05]
Statistical Analysis 2: Comparison: Panel B: MK-8266 BID, 1.8 mg vs Pooled Placebo; Test type: Other — Difference in change from baseline in cGMP; p = 0.17, Linear mixed effects model; Geometric Mean Ratio = 1.66, 90% CI 2-sided [0.66 to 4.17]
Statistical Analysis 3: Comparison: Panel C: MK-8266 TID, 1.8 mg vs Pooled Placebo; Test type: Other — Difference in change from baseline in cGMP; p = 0.054, Linear mixed effcts model; Geometric Mean Ratio = 0.41, 90% CI 2-sided [0.16 to 1.02]
Statistical Analysis 4: Comparison: Panels D & E Combined: MK-8266 TID, 2.4 mg vs Pooled Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Other — Difference in change from baseline in cGMP; p = 0.297, Linear mixed effcts model; Geometric Mean Ratio = 0.78, 90% CI 2-sided [0.35 to 1.73]

7. Secondary Outcome: Percent Inhibition of Platelet Aggregation Induced by Adenosine Diphosphate (ADP) Following Multiple Oral Doses of MK-8266 or Placebo
Description: The percent inhibition of ADP-induced platelet aggregation from Baseline to 5 hours postdose on Day 10 was assessed and is summarized here. Platelet aggregation was initiated by addition of ADP (2.5 µM) to the participant's blood sample. Aggregation was followed for 5 minutes after addition of the agonist, and the maximum percent of light transmission (extent of aggregation) obtained during this period, as well as the instrument-calculated slope (rate of aggregation), were reported. Post treatment platelet aggregation is expressed as a percent of each participant's pretreatment level of aggregation. Panel D and Panel E had identical treatments (MK-8266 0.8 mg TID), which were combined for this summary. The data are very limited. On Day 10 only 8 participants received MK-8266 0.8 mg TID and 3 participants received placebo.
Time Frame: Baseline and Day 10 (5 hours postdose)
Population: All participants who received at least one dose of the investigational drug and had assessment of ADP-induced platelet aggregation on Day 10
Measure: Mean (Standard Deviation); unit: Percent inhibition
Groups:
- Panels D & E Combined: MK-8266 TID (2.4 mg): MK-8266 0.8 mg TID, administered as oral capsules (2.4 mg) for 10 days. Panel D was completed prior to initiation of Panel E.
- Placebo: Matching placebo capsules, administered orally TID for 10 days
Arm/Group | Panels D & E Combined: MK-8266 TID (2.4 mg) | Placebo
Number analyzed (Participants) | 8 | 3
Percent inhibition | -12.3 (29.81) | -12.4 (18.89)

8. Secondary Outcome: Percent Inhibition of Platelet Aggregation Induced by Collagen Following Multiple Oral Doses of MK-8266 or Placebo
Description: The percent inhibition of collagen-induced platelet aggregation from Baseline to 5 hours postdose on Day 10 was assessed and is summarized here. Platelet aggregation was initiated by addition of collagen (2 µg/mL) to the participant's blood sample. Aggregation was followed for 5 minutes after addition of the agonist, and the maximum percent of light transmission (extent of aggregation) obtained during this period, as well as the instrument-calculated slope (rate of aggregation), were reported. Post treatment platelet aggregation is expressed as a percent of each participant's pretreatment level of aggregation. Panel D and Panel E had identical treatments (MK-8266 0.8 mg TID), which were combined for this summary. The data are very limited. On Day 10, only 8 participants received MK-8266 0.8 mg TID and 3 participants received placebo.
Time Frame: Baseline and Day 10 (5 hours postdose)
Population: All participants who received at least one dose of the investigational drug and had assessment of collagen-induced platelet aggregation on Day 10
Measure: Mean (Standard Deviation); unit: Percent inhibition
Arm/Group | Panels D & E Combined: MK-8266 TID (2.4 mg) | Placebo
Number analyzed (Participants) | 8 | 3
Percent inhibition | -17.7 (26.30) | -8.87 (33.76)

ADVERSE EVENTS:
Time Frame: 11 days
Groups:
- Panel A: Placebo BID; Panel B: Placebo BID: Matching placebo capsules, administered orally BID for 10 days
- Panel B: MK-8266 BID, 1.8 mg: MK-8266 1.8 mg (1 mg AM + 0.8 mg PM), administered orally for 10 days
- Panel D: MK-8266 TID, 2.4 mg; Panel E: MK-8266 TID, 2.4 mg: MK-8266 0.8 mg TID, administered as oral capsules (2.4 mg) for 10 days
Arm/Group | Panel A: MK-8266 BID, 1 mg | Panel A: Placebo BID | Panel B: MK-8266 BID, 1.8 mg | Panel B: Placebo BID | Panel C: MK-8266 TID, 1.8 mg | Panel C: Placebo TID | Panel D: MK-8266 TID, 2.4 mg | Panel D: Placebo TID | Panel E: MK-8266 TID, 2.4 mg | Panel E: Placebo TID
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2 | 0/6 | 0/2
Other Adverse Events (participants affected / at risk) | 5/6 | 0/2 | 5/6 | 1/2 | 3/6 | 1/2 | 4/6 | 1/2 | 5/6 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panel A: MK-8266 BID, 1 mg (N=6) | Panel A: Placebo BID (N=2) | Panel B: MK-8266 BID, 1.8 mg (N=6) | Panel B: Placebo BID (N=2) | Panel C: MK-8266 TID, 1.8 mg (N=6) | Panel C: Placebo TID (N=2) | Panel D: MK-8266 TID, 2.4 mg (N=6) | Panel D: Placebo TID (N=2) | Panel E: MK-8266 TID, 2.4 mg (N=6) | Panel E: Placebo TID (N=2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sluggishness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 4 (10) | 1 (1) | 3 (5) | 1 (1) | 2 (3) | 1 (3) | 4 (7) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.